CLINICAL TRIAL: NCT04939636
Title: The Influence of Vitamin D on the Physical Performance and General Health of Conscripts of the Estonian Defence Forces
Brief Title: Vitamin D Supplementation in Estonian Conscripts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tartu University Hospital (Other)
Collaborators: Estonian Defence Forces (Unknown); University of Tartu (Other)
Responsible Party: Principal Investigator, Leho Rips, Principal Investigator, MD, Orthopaedic surgeon, Tartu University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 323/T-3
Record Dates: First submitted 2020-10-13; First posted 2021-06-25 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Vitamin D Deficiency; Military Activity; Physical Stress
Keywords: Vitamin D supplementation; Conscripts; Military sevice; Physical preformance
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Triple blinded randomized placebo-controlled study
Who Masked: Participant, Care Provider, Investigator
Masking Description: Computed randomization will be used to divide conscripts into two groups; the intervention group, who received vitamin D3 capsules (4000 IU/100µg) or the intervention group, who received vitamin D3 capsules (600 IU/15µg)
  .
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D3 capsules 4000IU/100µg (Active Comparator): Get Vitamin D3 capsules 4000IU/100µg.
  Interventions: Dietary Supplement: Vitamin D3 capsules 4000IU/100µg.
- Vitamin D3 capsules 600IU/15µg (Active Comparator): Get Vitamin D3 capsules 600IU/15µg.
  Interventions: Dietary Supplement: Vitamin D3 capsules 600IU/15µg.

INTERVENTIONS:
Dietary Supplement: Vitamin D3 capsules 4000IU/100µg. — Vitamin D3 supplementation
  Arms: Vitamin D3 capsules 4000IU/100µg
Dietary Supplement: Vitamin D3 capsules 600IU/15µg. — Vitamin D3 supplementation
  Arms: Vitamin D3 capsules 600IU/15µg

SUMMARY:
A longitudinal, double-blinded, randomized, trial, with a 10 month follow-up period will be conducted between July 2021 to May 2022

DETAILED DESCRIPTION:
I DETAILED DESCRIPTION OF THE SUBJECTS AND THEIR RECRUITMENT Four hundred volunteers from the 2nd Infantry Brigade of the Kuperjanov Infantry Battalion (Võru, Estonia) aged 18-30 are invited to participate in this study. To this end, a general meeting will be held at the beginning of the conscription. The participants will be given an overview of the study, its objectives and methods, all the risks that may be involved, and the potential benefits. The meeting will emphasise the voluntary nature of the study and the fact that non-participation in the study does not lead to changes in the overall cost of their conscription. Conscripts wishing to participate in the study can sign an information sheet and informed consent form to participate in the study after the meeting. Based on previous studies (experience of our working group in 2014-2017), the participation of about 150-170 conscripts is expected (25-30% of the total number).

Places of the study:

1. University of Tartu Clinic, Sports Medicine and Rehabilitation Clinic, Sports Traumatology Centre, Puusepa 1a, Tartu, 51014
2. Recruitment of subjects, general medical assessment and completion of questionnaires, blood sampling, physical tests, and bone densitometry analysis. Kuperjanov Infantry Battalion, 2nd Infantry Brigade (Kose tee 3a, 65603, Võru)
3. Determination of vitamin D, PTH, and Ca in the blood: Synlab Eesti OÜ, Teguri 37b, 50107, Tartu

The questionnaires used in the study will be completed on site at the Kuperjanov Infantry Battalion. The subjects are divided into two groups by a computer with double-blind randomisation in a 1 : 1 ratio - subjects receiving 4,000 IU of vitamin D or a 100 µg capsule (Group I, n = 75-85) and subjects receiving 600 IU or 15 µg vitamin D capsules (Group II, n = 75-85) of the same shape and colour once a day with breakfast The corresponding capsules are pre-prepared in agreement with the manufacturer (HC CLOVER Productos y Servicios, S.Lk) and packed in standard jars (100 capsules per jar; a total of three jars with the corresponding number of capsules for ten months should be used for the study). Each jar is coded individually for each subject in accordance with the randomised groups.

Serum levels of vitamin D (25(OH)D), s-PTH, s-Ca, and s-iCa are determined in all subjects during the visits (SynLab Eesti OÜ, Tartu). Analyses are taken four times during the study (visits): July, October, February, and April/May. All analyses are determined at the end of the study at the same time to reduce intra-assay variability due to the use of different kits.

For all health-related problems related to the study, as well as other problems related to the study, conscripts are consulted by the orthopaedist in charge (Dr Leho Rips). If there are any health problems not related to the study, the medical staff of Kuperjanov will inform the principal researcher (Dr Leho Rips). The subjects have the right to contact the principal researcher directly in case of problems related to the study.

Exclusion from the study: - refusal of a conscript or withdrawal of consent, departure from military unit, force majeure, acute trauma, or illness in the course of conscript requiring hospital treatment. All these cases are recorded and taken into account in the subsequent analysis.

II DETAILED DESCRIPTION OF THE STUDY METHODOLOGY

Anthropometric measurements. The length of the body (LB) is measured with a metal anthropometer in a vertical position, the heels are together and the person measuring the subject ensures that the lower eyelid and the outer ear canal of the subject are in a horizontal plane. To determine body weight (W), the subject should wear as little clothes as possible. An electronic scale with a measuring accuracy of ± 0,1 kg is used for the measurement. The formula BMI = W / LB [kg/m2] is used to calculate the body mass index.

Vitamin D in serum ((25(OH)D is determined by chemiluminescence immunoassay (CLIA). (LIAISON 25 OH Vitamin D TOTAL Assay (REF 310600, DiaSorin Inc, USA)) with a sensitivity of 4 ng/ml and an intra-assay variability coefficient (CV) of 0.1-3.8%. Vitamin D levels in the blood are determined four times during the study period to explain the effects of strain, Estonian climate, and supplementation on serum concentrations (at the beginning of the conscript, twice in the middle of the conscript, and in the final phase).

Calcium (s-Ca), ionised calcium (s-iCa), and parathyroid hormone (s-PTH) are determined from blood serum by potentiometry and chemiluminescent immunoassay (CLIA), respectively.

All blood tests are taken at the same time in the morning before breakfast and during the same periods, analogously to vitamin D.

About 5 to 8 ml of blood is taken during each blood test, a total of 20 to 32 ml. This is about 2 tablespoons of blood throughout the study.

Assessment of knee pain. The visual analogue scale VAS is used where '0' - no pain and '10' - maximum pain, associated with the KOOS questionnaire to assess subjective complaints related to the knee joint.

Subjective assessment of knee joint function by the subject. The subjects evaluate the subjective complaints and function of the knee joint with a questionnaire (Knee Injury and Osteoarthritis Outcome Score, KOOS), which is used to find out their assessment of the condition of their knee(s) and how well they can cope with daily activities. It is possible to get a maximum of 100 points (no complaints) and a minimum of 0 points, which means extreme complaints.

Hand grip strength is determined by isometric contraction while standing, upper limb away from the body, using a hand dynamometer (Lafayette Instrument Co., USA). The studies use maximal hand grip strength as an indirect indicator of whole-body muscle strength.

Subjective assessment of physical activity by the subject. The Baecke Physical Activity Questionnaire consists of three parts and is based on a person's subjective assessment of their work, sport, and leisure (it is possible to get 1-5 points for each question). To interpret the results, the number of points in each subsection and the total number of points in the whole questionnaire are given. A similar questionnaire has been used to determine physical activity in previous studies in conscripts. IPAQ International Physical Activity Questionnaire, which assesses the level of physical activity in the last 7 days.

The assessment of subjective pain in different regions of the body is done with the Cornell Musculoskeletal Discomfort Questionnaires (CMDQ), where the intensity of pain and the region of the body can be noted. Pain questionnaire ( to assess pain in different regions of the body on a scale from 0 (none) to 10 (maximum possible pain).

The assessment of subjective health status and health-related quality of life by the subject is performed using standard questionnaires SF-36, RAND36, and BDI - Beck Depression Inventory. The questionnaires have been validated in Estonia and are valid for identifying health-related aspects. The questionnaires are based on the subject's assessment of their health aspects. The SF-36 questionnaire identifies the health status with a descriptive health profile and is more sensitive than other questionnaires. It also calculates the total physical and mental health scores. The BDI questionnaire is based on the assessment of the subject concerning aspects related to their mental health.

Evaluation of emotional well-being and somatic symptom disorder symptoms on the basis of the EEK-2 emotional well-being questionnaire and ACR 2010 questionnaires The emotional well-being questionnaire is a patient-completed self-assessment scale for identifying major depression and anxiety disorders and their adjacent symptoms in the past month. The EEK-2 questionnaire consists of 28 statements formulated based on diagnostic criteria and clinical feasibility. The answers are on a scale of 0-4 and the subject indicates how much the problem has disturbed them in the last month. The ACR 2010 questionnaire is a questionnaire developed and validated by the American College of Rheumatology to assess the presence of the somatic symptom disorder and non-physical pain (such as fibromyalgia) in subjects.

Fitness tests. Along with other data, the level of physical training of the conscripts is analysed using the standardised Army Physical Fitness Test (APFT), consisting of push-ups, sit-ups, and a 2-mile (3.2-km) run. The test has been adapted and used for a long time in the Estonian Defence Forces. Based on the results, the total score is calculated.

Bone density study or densitometry. A mobile DXL machine is used to determine bone density. Bone density is determined from the heel bone. Bone density is determined twice during the study period on site. Bone density measurement of the heel bone is performed by densitometry with a DXL Calscan instrument (Demetech AB, SWE). The measurements are performed at the beginning of the study and after about 10 months, just before the end of the conscript. The procedure shows the bone density of the subjects. The second study provides an assessment of the effects of exercise on the musculoskeletal system.

Health status monitoring. The health status of conscripts is monitored in the medical centre of the Combat Service Support Battalion of the 2nd Infantry Brigade, where records are made of the appeals and complaints of the conscripts, the number of days in inpatient care and bed rest, and the number of days when a conscript was absent from the conscript due to health problems.

Evaluation of vitamin D content in food rations of the Defence Forces. The average daily vitamin D content of the 1-month period of conscription in the daily food ration for conscripts is assessed. Based on international analytical data on vitamin D content in food.

Questionnaire completion and data collection, blood sampling, anthropometric evaluations, and health monitoring are performed by the study team.

ELIGIBILITY:
Inclusion Criteria:

1. Participating in military service at the Estonian Defence Forces
2. Voluntary participation in the study

Exclusion Criteria:

1. Refusal of a conscript or withdrawal of consent
2. Departure from military unit
3. Force majeure
4. Acute trauma or illness in the course of conscript requiring hospital treatment
5. Serious side effects or allergies to vitamin D capsules

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2021-07-19 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2022-06-16 (Actual)

PRIMARY OUTCOMES:
Prevalence of vitamin D between study groups (Baseline, no intervention) | 0 months Baseline
  Prevalence of vitamin D measured serum vitamin D 25(OH)D concentration. Vitamin D considered as sufficient if the serum 25(OH)D concentration is ≥75 nmol/L, insufficient if <75 nmol/L, deficient if <50 nmol/L and critical deficiency < 25 nmol/L.
Prevalence of vitamin D between study groups (Intervention I vs.II) | 3 months
  Prevalence of vitamin D measured serum vitamin D 25(OH)D concentration. Vitamin D considered as sufficient if the serum 25(OH)D concentration is ≥75 nmol/L, insufficient if <75 nmol/L, deficient if <50 nmol/L and critical deficiency < 25 nmol/L.
Prevalence of vitamin D between study groups (Intervention I vs.II) | app.6-7 months
  Prevalence of vitamin D measured serum vitamin D 25(OH)D concentration. Vitamin D considered as sufficient if the serum 25(OH)D concentration is ≥75 nmol/L, insufficient if <75 nmol/L, deficient if <50 nmol/L and critical deficiency < 25 nmol/L.
Prevalence of vitamin D between study groups (Intervention I vs.II) | app. 9-10 months
  Prevalence of vitamin D measured serum vitamin D 25(OH)D concentration. Vitamin D considered as sufficient if the serum 25(OH)D concentration is ≥75 nmol/L, insufficient if <75 nmol/L, deficient if <50 nmol/L and critical deficiency < 25 nmol/L.

SECONDARY OUTCOMES:
Serum parathyroid hormone | 0 months baseline
  Serum parathyroid hormone concentration (pmol/l)
Serum parathyroid hormone | 3 months
  Serum parathyroid hormone concentration (pmol/l)
Serum parathyroid hormone | app. 6-7 months
  Serum parathyroid hormone concentration (pmol/l)
Serum parathyroid hormone | app. 9-10 months
  Serum parathyroid hormone concentration (pmol/l)
Serum calcium | 0 months baseline
  Serum calcium (Ca) concentration (mmol/l)
Serum calcium | 3 months
  Serum calcium (Ca) concentration (mmol/l)
Serum calcium | app.6-7 months
  Serum calcium (Ca) concentration (mmol/l)
Serum calcium | app. 9-10 months
  Serum calcium (Ca) concentration (mmol/l)
Serum ionized calcium | 0 months baseline
  Serum ionized calcium (Ca-i) concentration (mmol/l)
Serum ionized calcium | app. 3 months
  Serum ionized calcium (Ca-i) concentration (mmol/l)
Serum ionized calcium | app.6-7 months
  Serum ionized calcium (Ca-i) concentration (mmol/l)
Serum ionized calcium | app.9-10 months
  Serum ionized calcium (Ca-i) concentration (mmol/l)
Knee pain The visual analogue scale VAS | 0 months baseline
  To assess subjective complaints related to the knee joint. The visual analogue scale VAS is used where '0' - no pain and '10' - maximum pain
Knee pain The visual analogue scale VAS | 3 months
  To assess subjective complaints related to the knee joint. The visual analogue scale VAS is used where '0' - no pain and '10' - maximum pain
Knee pain The visual analogue scale VAS | app. 6-7 months
  To assess subjective complaints related to the knee joint. The visual analogue scale VAS is used where '0' - no pain and '10' - maximum pain
Knee pain The visual analogue scale VAS | app.9-10 months
  To assess subjective complaints related to the knee joint. The visual analogue scale VAS is used where '0' - no pain and '10' - maximum pain
Subjective assessment of knee joint function KOOS | 0 months baseline
  The subjects evaluate the subjective complaints and function of the knee joint with a questionnaire. It is possible to get a maximum of 100 points (no complaints) and a minimum of 0 points, which means extreme complaints.
Subjective assessment of knee joint function KOOS | 3 months
  The subjects evaluate the subjective complaints and function of the knee joint with a questionnaire. It is possible to get a maximum of 100 points (no complaints) and a minimum of 0 points, which means extreme complaints.
Subjective assessment of knee joint function KOOS | app. 6-7 months
  The subjects evaluate the subjective complaints and function of the knee joint with a questionnaire. It is possible to get a maximum of 100 points (no complaints) and a minimum of 0 points, which means extreme complaints.
Subjective assessment of knee joint function KOOS | app. 9-10 months
  The subjects evaluate the subjective complaints and function of the knee joint with a questionnaire. It is possible to get a maximum of 100 points (no complaints) and a minimum of 0 points, which means extreme complaints.
Hand grip strength | 0 months baseline
  Is determined by isometric contraction while standing, upper limb away from the body, using a hand dynamometer (Lafayette Instrument Co., USA)
Hand grip strength | 3 months
  Is determined by isometric contraction while standing, upper limb away from the body, using a hand dynamometer (Lafayette Instrument Co., USA)
Hand grip strength | app.6-7 months
  Is determined by isometric contraction while standing, upper limb away from the body, using a hand dynamometer (Lafayette Instrument Co., USA)
Hand grip strength | app.9-10 months
  Is determined by isometric contraction while standing, upper limb away from the body, using a hand dynamometer (Lafayette Instrument Co., USA)
Subjective assessment of physical activity by the subject (Baeckley). | 0 months baseline
  The Baecke Physical Activity Questionnaire consists of three parts and is based on a person's subjective assessment of their work, sport, and leisure. Each domain could receive a score from one to five points, thus allowing a total score from three (minimum) to fifteen (maximum).
Subjective assessment of physical activity by the subject (IPAQ). | 0 months baseline
  International Physical Activity Questionnaire, which assesses the level of physical activity in the last 7 days. Categorical Score- three levels of physical activity are presented - low, medium and high.
Subjective assessment of physical activity by the subject (IPAQ). | 3 months
  International Physical Activity Questionnaire, which assesses the level of physical activity in the last 7 days. Categorical Score- three levels of physical activity are presented - low, medium and high.
Subjective assessment of physical activity by the subject (IPAQ). | app. 6-7 months
  International Physical Activity Questionnaire, which assesses the level of physical activity in the last 7 days. Categorical Score- three levels of physical activity are presented - low, medium and high.
Subjective assessment of physical activity by the subject (IPAQ). | app. 9-10 months
  International Physical Activity Questionnaire, which assesses the level of physical activity in the last 7 days. Categorical Score- three levels of physical activity are presented - low, medium and high.
The assessment of subjective pain in different regions of the body (Cornell) | 0 months baseline
  Is done with the Cornell Musculoskeletal Discomfort Questionnaires where the intensity of pain and the region of the body can be noted as 'mild', 'moderate' and 'severe discomfort'.
The assessment of subjective pain in different regions of the body (Cornell) | 3 months
  Is done with the Cornell Musculoskeletal Discomfort Questionnaires where the intensity of pain and the region of the body can be noted as 'mild', 'moderate' and 'severe discomfort'
The assessment of subjective pain in different regions of the body (Cornell) | app. 6-7 months
  Is done with the Cornell Musculoskeletal Discomfort Questionnaires where the intensity of pain and the region of the body can be noted as 'mild', 'moderate' and 'severe discomfort'.
The assessment of subjective pain in different regions of the body (Cornell) | app.9-10 months
  Is done with the Cornell Musculoskeletal Discomfort Questionnaires where the intensity of pain and the region of the body can be noted as 'mild', 'moderate' and 'severe discomfort'.
Pain questionnaire | 0 months baseline
  To assess pain in different regions of the body on a scale from 0 (none) to 10 (maximum possible pain)
Pain questionnaire | 3 months
  To assess pain in different regions of the body on a scale from 0 (none) to 10 (maximum possible pain)
Pain questionnaire | app. 6-7 months
  To assess pain in different regions of the body on a scale from 0 (none) to 10 (maximum possible pain)
Pain questionnaire | app. 9-10 months
  To assess pain in different regions of the body on a scale from 0 (none) to 10 (maximum possible pain)
The assessment of subjective health status and health-related quality of life by the subject-RAND-36. | 0 months baseline
  Is performed using standard questionnaires RAND 36. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.
The assessment of subjective health status and health-related quality of life by the subject- RAND-36. | 3 months
  Is performed using standard questionnaires RAND 36. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.
The assessment of subjective health status and health-related quality of life by the subject- RAND-36. | app.6-7 months
  Is performed using standard questionnaires RAND 36. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.
The assessment of subjective health status and health-related quality of life by the subject- RAND 36. | app.9-10 months
  Is performed using standard questionnaires RAND 36. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.
The assessment of subjective health status and health-related quality of life by the subject - Beck Depression | 0 months - baselilne
  Is performed using standard questionnaires - Beck Depression Inventory. The BDI questionnaire is based on the assessment of the subject concerning aspects related to their mental health. Total score of 0-13 is considered minimal range, 14-19 is mild, 20-28 is moderate, and 29-63 is severe depression.
The assessment of subjective health status and health-related quality of life by the subject - Beck Depression | 3 months
  Is performed using standard questionnaires - Beck Depression Inventory. The BDI questionnaire is based on the assessment of the subject concerning aspects related to their mental health. Total score of 0-13 is considered minimal range, 14-19 is mild, 20-28 is moderate, and 29-63 is severe depression.
The assessment of subjective health status and health-related quality of life by the subject - Beck Depression | app. 6-7 months
  Is performed using standard questionnaires - Beck Depression Inventory. The BDI questionnaire is based on the assessment of the subject concerning aspects related to their mental health. Total score of 0-13 is considered minimal range, 14-19 is mild, 20-28 is moderate, and 29-63 is severe depression.
The assessment of subjective health status and health-related quality of life by the subject - Beck Depression | app. 9-10 months
  Is performed using standard questionnaires - Beck Depression Inventory. The BDI questionnaire is based on the assessment of the subject concerning aspects related to their mental health. Total score of 0-13 is considered minimal range, 14-19 is mild, 20-28 is moderate, and 29-63 is severe depression.
Evaluation of emotional well-being and somatic symptom disorder symptoms - EEK-2 | 0 months baseline
  On the basis of the EEK-2 emotional well-being questionnaire. The emotional well-being questionnaire is a patient-completed self-assessment scale for identifying major depression and anxiety disorders and their adjacent symptoms in the past month. The EEK-2 questionnaire consists of 28 statements formulated based on diagnostic criteria and clinical feasibility. The answers are on a scale of 0-4 and the subject indicates how much the problem has disturbed them in the last month.
Evaluation of emotional well-being and somatic symptom disorder symptoms - EEK-2 | 3 months baseline
  On the basis of the EEK-2 emotional well-being questionnaire.The emotional well-being questionnaire is a patient-completed self-assessment scale for identifying major depression and anxiety disorders and their adjacent symptoms in the past month. The EEK-2 questionnaire consists of 28 statements formulated based on diagnostic criteria and clinical feasibility. The answers are on a scale of 0-4 and the subject indicates how much the problem has disturbed them in the last month.
Evaluation of emotional well-being and somatic symptom disorder symptoms- EEK-2. | app. 6-7 months
  On the basis of the EEK-2 emotional well-being questionnaire.The emotional well-being questionnaire is a patient-completed self-assessment scale for identifying major depression and anxiety disorders and their adjacent symptoms in the past month. The EEK-2 questionnaire consists of 28 statements formulated based on diagnostic criteria and clinical feasibility. The answers are on a scale of 0-4 and the subject indicates how much the problem has disturbed them in the last month.
Evaluation of emotional well-being and somatic symptom disorder symptoms -EEK-2 | app.9-10 months
  On the basis of the EEK-2 emotional well-being questionnaire.The emotional well-being questionnaire is a patient-completed self-assessment scale for identifying major depression and anxiety disorders and their adjacent symptoms in the past month. The EEK-2 questionnaire consists of 28 statements formulated based on diagnostic criteria and clinical feasibility. The answers are on a scale of 0-4 and the subject indicates how much the problem has disturbed them in the last month.
Evaluation of emotional well-being and somatic symptom disorder symptoms - ACR 2010 | 0 months - baseline
  The ACR 2010 questionnaire is a questionnaire developed and validated by the American College of Rheumatology to assess the presence of the somatic symptom disorder and non-physical pain (such as fibromyalgia) in subjects. Pain score 0 no pain and 19 maximum pain. Symptoms score 0 - no symptoms and 12 maximum symptoms.
Evaluation of emotional well-being and somatic symptom disorder symptoms ACR 2010 | 3 months
  The ACR 2010 questionnaire is a questionnaire developed and validated by the American College of Rheumatology to assess the presence of the somatic symptom disorder and non-physical pain (such as fibromyalgia) in subjects. Pain score 0 no pain and 19 maximum pain. Symptoms score 0 - no symptoms and 12 maximum symptoms.
Evaluation of emotional well-being and somatic symptom disorder symptoms ACR 2010 | app. 6-7 months
  The ACR 2010 questionnaire is a questionnaire developed and validated by the American College of Rheumatology to assess the presence of the somatic symptom disorder and non-physical pain (such as fibromyalgia) in subjects. Pain score 0 no pain and 19 maximum pain. Symptoms score 0 - no symptoms and 12 maximum symptoms.
Evaluation of emotional well-being and somatic symptom disorder symptoms ACR 2010 | app. 9-10 months
  The ACR 2010 questionnaire is a questionnaire developed and validated by the American College of Rheumatology to assess the presence of the somatic symptom disorder and non-physical pain (such as fibromyalgia) in subjects. Pain score 0 no pain and 19 maximum pain. Symptoms score 0 - no symptoms and 12 maximum symptoms.
Fitness tests | 0 months baseline
  the level of physical training of the conscripts is analysed using the standardised Army Physical Fitness Test (APFT). Soldiers were scored based on their performance in three events consisting of the push-up, sit-up, and a two-mile run, ranging from 0 to 100 points in each event. A minimum score of 60 in each event was required to pass the test. The soldier's overall score was the sum of the points from the three events. If a soldier passed all three events, the total could have range from 180 to 300.
Fitness tests | app 5 months
  the level of physical training of the conscripts is analysed using the standardised Army Physical Fitness Test (APFT). Soldiers were scored based on their performance in three events consisting of the push-up, sit-up, and a two-mile run, ranging from 0 to 100 points in each event. A minimum score of 60 in each event was required to pass the test. The soldier's overall score was the sum of the points from the three events. If a soldier passed all three events, the total could have range from 180 to 300.
Fitness tests | app 9-10 months
  the level of physical training of the conscripts is analysed using the standardised Army Physical Fitness Test (APFT). Soldiers were scored based on their performance in three events consisting of the push-up, sit-up, and a two-mile run, ranging from 0 to 100 points in each event. A minimum score of 60 in each event was required to pass the test. The soldier's overall score was the sum of the points from the three events. If a soldier passed all three events, the total could have range from 180 to 300.
Bone density study or densitometry | 0 months baseline
  A mobile DXL machine is used to determine bone density
Bone density study or densitometry | app.9-10 months
  A mobile DXL machine is used to determine bone density
Health status monitoring - upper respiratory tract infections (UTRI) | During all the study (daily 0-10 months)
  The health status of conscripts is monitored in the medical centre of the Combat Service Support Battalion of the 2nd Infantry Brigade, where records are made of the appeals and complaints of the conscripts, the number of days in inpatient care and bed rest, and the number of days when a conscript was absent from the conscript due to upper respiratory infection (UTRI).
Health status monitoring - musculoskeletal injury | During all the study (daily 0-10 months)
  The health status of conscripts is monitored in the medical centre of the Combat Service Support Battalion of the 2nd Infantry Brigade, where records are made of the appeals and complaints of the conscripts, the number of days in inpatient care and bed rest, and the number of days when a conscript was absent from the conscript due to musculoskeletal injury.
Bone density study or densitometry | app. 6 months
  A mobile DXL machine is used to determine bone density

CONTACTS AND LOCATIONS:
Overall Officials: Madis Rahu, PhD, Study Director — University of Tartu
Locations (1):
- Kuperjanov Infantry Battalion, Estonian Defence Forces, Võru, Võrumaa, Estonia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baecke JA, Burema J, Frijters JE. A short questionnaire for the measurement of habitual physical activity in epidemiological studies. Am J Clin Nutr. 1982 Nov;36(5):936-42. doi: 10.1093/ajcn/36.5.936. PMID 7137077
- [Background] Bischoff-Ferrari HA, Giovannucci E, Willett WC, Dietrich T, Dawson-Hughes B. Estimation of optimal serum concentrations of 25-hydroxyvitamin D for multiple health outcomes. Am J Clin Nutr. 2006 Jul;84(1):18-28. doi: 10.1093/ajcn/84.1.18. PMID 16825677
- [Background] Dawson-Hughes B, Heaney RP, Holick MF, Lips P, Meunier PJ, Vieth R. Estimates of optimal vitamin D status. Osteoporos Int. 2005 Jul;16(7):713-6. doi: 10.1007/s00198-005-1867-7. Epub 2005 Mar 18. PMID 15776217
- [Background] EFSA Panel on Dietetic Products, Nutrition and Allergies (NDA); Turck D, Bresson JL, Burlingame B, Dean T, Fairweather-Tait S, Heinonen M, Hirsch-Ernst KI, Mangelsdorf I, McArdle HJ, Naska A, Nowicka G, Pentieva K, Sanz Y, Siani A, Sjodin A, Stern M, Tome D, Van Loveren H, Vinceti M, Willatts P, Lamberg-Allardt C, Przyrembel H, Tetens I, Dumas C, Fabiani L, Ioannidou S, Neuhauser-Berthold M. Dietary reference values for vitamin K. EFSA J. 2017 May 22;15(5):e04780. doi: 10.2903/j.efsa.2017.4780. eCollection 2017 May. PMID 32625486
- [Background] Goodman GP, Schoenfeld AJ, Owens BD, Dutton JR, Burks R, Belmont PJ. Non-emergent orthopaedic injuries sustained by soldiers in Operation Iraqi Freedom. J Bone Joint Surg Am. 2012 Apr 18;94(8):728-35. doi: 10.2106/JBJS.K.00129. PMID 22517389
- [Background] Hughes JM, Smith MA, Henning PC, Scofield DE, Spiering BA, Staab JS, Hydren JR, Nindl BC, Matheny RW Jr. Bone formation is suppressed with multi-stressor military training. Eur J Appl Physiol. 2014 Nov;114(11):2251-9. doi: 10.1007/s00421-014-2950-6. Epub 2014 Jul 16. PMID 25027064
- [Background] Hypponen E, Power C. Hypovitaminosis D in British adults at age 45 y: nationwide cohort study of dietary and lifestyle predictors. Am J Clin Nutr. 2007 Mar;85(3):860-8. doi: 10.1093/ajcn/85.3.860. PMID 17344510
- [Background] Inklebarger J, Griffin M, Taylor MJ, Dembry RB. Femoral and tibial stress fractures associated with vitamin D insufficiency. J R Army Med Corps. 2014 Mar;160(1):61-3. doi: 10.1136/jramc-2013-000085. Epub 2013 Jun 26. PMID 24109098
- [Background] Knapik JJ, East WB. History of United States Army physical fitness and physical readiness training. US Army Med Dep J. 2014 Apr-Jun:5-19. PMID 24706237
- [Background] Kull M Jr, Kallikorm R, Tamm A, Lember M. Seasonal variance of 25-(OH) vitamin D in the general population of Estonia, a Northern European country. BMC Public Health. 2009 Jan 19;9:22. doi: 10.1186/1471-2458-9-22. PMID 19152676
- [Background] Laaksi IT, Ruohola JP, Ylikomi TJ, Auvinen A, Haataja RI, Pihlajamaki HK, Tuohimaa PJ. Vitamin D fortification as public health policy: significant improvement in vitamin D status in young Finnish men. Eur J Clin Nutr. 2006 Aug;60(8):1035-8. doi: 10.1038/sj.ejcn.1602414. Epub 2006 Feb 15. PMID 16482069
- [Background] Laaksi I, Ruohola JP, Tuohimaa P, Auvinen A, Haataja R, Pihlajamaki H, Ylikomi T. An association of serum vitamin D concentrations < 40 nmol/L with acute respiratory tract infection in young Finnish men. Am J Clin Nutr. 2007 Sep;86(3):714-7. doi: 10.1093/ajcn/86.3.714. PMID 17823437
- [Background] Laaksi I, Ruohola JP, Mattila V, Auvinen A, Ylikomi T, Pihlajamaki H. Vitamin D supplementation for the prevention of acute respiratory tract infection: a randomized, double-blinded trial among young Finnish men. J Infect Dis. 2010 Sep 1;202(5):809-14. doi: 10.1086/654881. No abstract available. PMID 20632889
- [Background] Li-Ng M, Aloia JF, Pollack S, Cunha BA, Mikhail M, Yeh J, Berbari N. A randomized controlled trial of vitamin D3 supplementation for the prevention of symptomatic upper respiratory tract infections. Epidemiol Infect. 2009 Oct;137(10):1396-404. doi: 10.1017/S0950268809002404. Epub 2009 Mar 19. PMID 19296870
- [Background] Maloney SR, Almarines D, Goolkasian P. Vitamin D levels and monospot tests in military personnel with acute pharyngitis: a retrospective chart review. PLoS One. 2014 Jul 10;9(7):e101180. doi: 10.1371/journal.pone.0101180. eCollection 2014. PMID 25009977
- [Background] Ong GS, Walsh JP, Stuckey BG, Brown SJ, Rossi E, Ng JL, Nguyen HH, Kent GN, Lim EM. The importance of measuring ionized calcium in characterizing calcium status and diagnosing primary hyperparathyroidism. J Clin Endocrinol Metab. 2012 Sep;97(9):3138-45. doi: 10.1210/jc.2012-1429. Epub 2012 Jun 28. PMID 22745247
- [Background] Ruohola JP, Laaksi I, Ylikomi T, Haataja R, Mattila VM, Sahi T, Tuohimaa P, Pihlajamaki H. Association between serum 25(OH)D concentrations and bone stress fractures in Finnish young men. J Bone Miner Res. 2006 Sep;21(9):1483-8. doi: 10.1359/jbmr.060607. PMID 16939407
- [Background] Wierniuk A, Wlodarek D. Estimation of energy and nutritional intake of young men practicing aerobic sports. Rocz Panstw Zakl Hig. 2013;64(2):143-8. PMID 23987084